CLINICAL TRIAL: NCT07378644
Title: A Phase 2/3 Randomized, Double Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Pharmacodynamics, Safety and Efficacy of SKY-0515 in Participants With Huntington's Disease
Brief Title: Study to Evaluate the Pharmacodynamics, Safety and Efficacy of SKY-0515 in Participants With Huntington's Disease
Acronym: FALCON-HD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Skyhawk Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKY-0515-004-WW
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Huntington Disease
Keywords: SKY-0515; Skyhawk; HTT; Neurodegenerative; Huntington Disease; mRNA; Splicing; Mutant Huntingtin protein
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled dose ranging
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator (1) (Active Comparator): Dosage Level(s): Low Dose
  Interventions: Drug: SKY-0515
- Active Comparator (2) (Active Comparator): Dosage Level(s): Mid Dose
  Interventions: Drug: SKY-0515
- Active Comparator (3) (Active Comparator): Dosage Level(s): High Dose
  Interventions: Drug: SKY-0515
- Placebo Comparator (4) (Placebo Comparator): Matching placebo once daily oral
  Interventions: Drug: SKY-0515 Placebo

INTERVENTIONS:
Drug: SKY-0515 — Type: Small molecule Dosage Level(s): Low, mid, high Route of Administration: Oral Dosage Frequency: Once daily Blinded Treatment Duration: 18 months Use: Experimental
  Arms: Active Comparator (1); Active Comparator (2); Active Comparator (3)
Drug: SKY-0515 Placebo — Route of Administration: Oral Dosage Frequency: Once daily Blinded Treatment Duration: 18 months Use: Experimental
  Arms: Placebo Comparator (4)

SUMMARY:
The goal of this clinical trial is to test if the drug SKY-0515, an oral medication, can lower harmful proteins linked to Huntington's Disease (HD) and improve the symptoms of participants with HD. This study includes men and women aged 25 and older who have HD confirmed by genetic testing and meet certain requirements for physical ability and independence.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled trial conducted across multiple sites. This clinical trial aims to evaluate the safety, pharmacodynamics, and efficacy of SKY-0515, a novel, orally administered small molecule. Huntington's Disease (HD) is a rare, inherited neurodegenerative condition caused by a mutation in the huntingtin (HTT) gene, resulting in excessive production of mutant huntingtin (mHTT) protein, which damages nerve cells and leads to progressive motor, cognitive, and psychiatric symptoms. SKY-0515 is designed to reduce mHTT protein levels, leading to a decrease in both wild-type and mutant forms of HTT protein. Additionally, the drug lowers postmeiotic segregation 1 (PMS1) protein, which plays a role in somatic CAG repeat expansion-a key driver of HD progression. Participants must be aged 25 or older, have genetically confirmed HD (CAG repeat length ≥ 40), and meet specific functional and motor criteria. They will be assigned randomly to one of four treatment arms (three doses of SKY-0515 and one placebo group). Safety and efficacy will be evaluated through blood tests, imaging (MRI), and clinical assessments, including the Unified Huntington's Disease Rating Scale (UHDRS).

ELIGIBILITY:
Inclusion Criteria:

* 25 years or older.
* Huntington's Disease confirmed through genetic testing, with a specific change in exon 1 of the HTT gene (CAG repeat of 40 or more).
* Total Functional Capacity (TFC) score of 10 or more).
* Total Motor Score (TMS) of 6 or more).
* Independence Score (IS) of 70 or more).
* Women who can have children must have a negative pregnancy test before starting and use two types of birth control during the study and for 30 days after the last dose of the study drug.
* Men must agree to use birth control during the study and for 90 days after the last dose.
* Agree to sign a consent form and follow the study's rules and schedule.

Exclusion Criteria:

* Other Serious health problems or brain/spinal issues that could interfere with the study or make procedures unsafe.
* Conditions that interfere with protocol-specified assessments, like an implanted medical device or difficulty getting an MRI.
* Cancer, except for some types of skin cancer, or a history of cancer in the last five years.
* Severe allergies or have reacted badly to similar drugs in the past.
* Taking medications or treatments that might interfere with the study.
* Participated in another study or taken experimental drugs in the last two months (or longer for some drugs).
* Any kind of gene therapy.
* History of suicidal thoughts, severe depression, or have attempted suicide in the past year.
* Liver function tests show significant abnormalities.
* Positive for hepatitis B, hepatitis C, or HIV.
* Pregnancy, breastfeeding, or planning to become pregnant during the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Z-score from the Composite Unified Huntington's Disease Rating Scale (cUHDRS) | 72 weeks
  cUHDRS includes the Total Functional Capacity (range, 0-13; higher score means better functioning), Total Motor Score (range, 0-124; higher score means worse motor severity), Symbol Digit Modality Test (range, 0-110, correctly paired numbers-symbols in 90 seconds; higher score means better cognitive performance), and Stroop Color and Word Test (range, 0-no max value, correctly read color words in 45 seconds; higher score means better cognitive performance) scores. A z-score for each test is calculated, which alone can be used to describe relationship between an individual's test score and the mean score of a target population. A z-score of 0 is the mean, and ±1 is 1 standard deviation from the mean. For cUHDRS, z-scores of each test are summed, whereby a higher cUHDRS score is better (score of -3.06-no max value) and a change of ≥1.2 is a meaningful worsening, shown to track functional decline.

SECONDARY OUTCOMES:
Change from Baseline in Total Motor Score (TMS) | 72 weeks
  The total motor score (TMS) assessed motor features of HD with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural stability. Some items (such as chorea and dystonia) required grading each extremity (face, bucco-oral-lingual, and trunk) separately. Eye movements require both horizontal and vertical grades. The total motor impairment score is the sum of all the individual 31 motor sub-items (each rated from 0 to 4), with higher scores indicating more severe motor impairment than lower scores. The range of TMS is 0-124.
Change from Baseline in Total Functional Capacity (TFC) | 72 weeks
  TFC consists of five ordinally scaled items assessing a person's capacity with: (1) occupation; (2) financial affairs; (3) domestic responsibilities; (4) activities of daily living; and (5) independent living. Total score ranges from zero (worst) to 13 (best).
Change from Baseline in Independence Scale Score (IS) | 72 weeks
  The independence scale assesses independence on a 0 to 100 scale with higher scores indicating better functioning.
Change from Baseline in Symbol Digit Modalities Test (SDMT) | 72 weeks
  The SDMT assesses attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed. The score is the number of correctly paired abstract symbols and specific numbers in 90 seconds with higher scores indicating better cognitive functioning.
Change from Baseline in the Stroop Color and Word Test (SCWT) | 72 weeks
  In the Stroop Color and Word Test (SCWT) the number of words and colors read correctly is counted, with a higher score indicating better cognitive performance scores. There is no upper limit for SWR as it is a time-based task. The lower limit (worst possible) however is 0; higher score is better meaning less severity.

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Pineo Medical Ecosystem, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Skyhawk Therapeutics Website — https://www.skyhawktx.com/